CLINICAL TRIAL: NCT04617613
Title: Comparing Different Regimens for Eradication of Helicobacter Pylori in Kuwait
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Mohamed Alboraie, Postgraduate clinical researcher, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MKH-01-2016
Record Dates: First submitted 2020-10-29; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Omeprazole; Amoxicillin; Metronidazole; Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard triple therapy (Active Comparator): Standard triple therapy group received omeprazole 20 mg, amoxicillin 1 g and clarithromycin 500 mg twice daily for 14 days.
  Interventions: Drug: Omeprazole, Amoxicillin and Clarithromycin
- Quadruple therapy group (Experimental): Quadruple therapy group received omeprazole 20 mg, amoxicillin 1 g, clarithromycin 500 mg, and metronidazole 500 mg twice daily after meals for 14 days.
  Interventions: Drug: Omeprazole, Amoxicillin, Metronidazole and Clarithromycin

INTERVENTIONS:
Drug: Omeprazole, Amoxicillin, Metronidazole and Clarithromycin — The first group (standard triple therapy group) received omeprazole 20 mg, amoxicillin 1 g and clarithromycin 500 mg. The second group (quadruple therapy group) received omeprazole 20 mg, amoxicillin 1 g, clarithromycin 500 mg, and metronidazole 500 mg. Patients in both groups received omeprazole capsule twice daily before meals and the rest of the drugs twice daily after meals for 14 days.
  Other Names: Quadruple therapy group
  Arms: Quadruple therapy group
Drug: Omeprazole, Amoxicillin and Clarithromycin — The first group (standard triple therapy group) received omeprazole 20 mg, amoxicillin 1 g and clarithromycin 500 mg. The second group (quadruple therapy group) received omeprazole 20 mg, amoxicillin 1 g, clarithromycin 500 mg, and metronidazole 500 mg. Patients in both groups received omeprazole capsule twice daily before meals and the rest of the drugs twice daily after meals for 14 days.
  Other Names: Standard triple therapy
  Arms: Standard triple therapy

SUMMARY:
Eradication of H. pylori reduces morbidity in patients with chronic gastritis and can prevent gastric cancer. We aimed to evaluate the efficacy of clarithromycin-based triple therapy and non-bismuth based quadruple therapy for eradicating H. pylori in patients with chronic gastritis in Kuwait.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) induced chronic infection is associated with peptic ulcer, chronic gastritis, gastric cancer, and increasing antibiotic resistance. Eradication of H. pylori reduces morbidity in patients with chronic gastritis and can prevent gastric cancer in the high-risk population. We aimed to evaluate the efficacy of clarithromycin-based triple therapy and non-bismuth based quadruple therapy for eradicating H. pylori in patients with chronic gastritis in Kuwait. We enrolled treatment-naive dyspeptic patients with gastric biopsy-proven chronic gastritis secondary to H. pylori in a prospective, open-label, randomized study conducted at the gastroenterology outpatient clinics of Haya Habeeb gastroenterology center in Kuwait. Patients were randomized into two groups: the first group received the standard triple therapy (omeprazole, amoxicillin, and clarithromycin) for 14 days; and the second group received quadruple therapy (omeprazole, amoxicillin, clarithromycin, and metronidazole) for 14 days. All patients were tested for the eradication of H. pylori by carbon-13 urea breath test (13C-UBT) one month after completion of eradication therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female dyspeptic subjects aged ≥18 years with any nationality
* Patients with gastric biopsy-proven H. pylori related chronic gastritis and no other abnormalities in the upper gastrointestinal tract upon endoscopy
* Patients who were naive to treatment for H. pylori infection.

Exclusion Criteria:

* Pregnant or breastfeeding females
* Patients who were previously treated for H. pylori infection
* Patients who received any antibiotics, bismuth or acid-suppressant drugs within the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Negative 13-Carbon urea breath test | One month
  H. pylori eradication rate defined as negative 13-Carbon urea breath test (13C-UBT) one month after treatment
Adverse events | One month
  Any reported adverse events during the study period

REFERENCES:
- [Derived] Alfadhli A, Alboraie M, Afifi M, Dangi A. A Randomized Clinical Trial Comparing Triple Therapy versus Non-bismuth based Quadruple Therapy for the Eradication of Helicobacter Pylori in Kuwait. J Glob Infect Dis. 2022 Aug 26;14(3):99-105. doi: 10.4103/jgid.jgid_13_22. eCollection 2022 Jul-Sep. PMID 36237565